CLINICAL TRIAL: NCT00024063
Title: A Phase I Study Of SU006668 Via Twice Daily Oral Administration Under Fed Conditions In Patients With Advanced Malignancies
Brief Title: SU006668 in Treating Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068888; UCLA-0004061; SUGEN-SU6668.004; NCI-G01-2010
Record Dates: First submitted 2001-09-13; First posted 2004-04-06 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2007-04

CONDITIONS: Breast Cancer; Colorectal Cancer; Gastric Cancer; Kidney Cancer; Lung Cancer; Multiple Myeloma and Plasma Cell Neoplasm; Pancreatic Cancer; Prostate Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; stage IIIB breast cancer; recurrent non-small cell lung cancer; stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; refractory multiple myeloma; stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer; stage III multiple myeloma; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; male breast cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Kidney Neoplasms; Lung Neoplasms; Multiple Myeloma; Neoplasms, Plasma Cell; Pancreatic Neoplasms; Prostatic Neoplasms; Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung; Rectal Neoplasms; Carcinoma, Renal Cell; Breast Neoplasms, Male | interventions — orantinib

INTERVENTIONS:
Drug: orantinib

SUMMARY:
RATIONALE: Drugs such as SU006668 may stop the growth of solid tumors by stopping blood flow to the tumor.

PURPOSE: Phase I trial to study the effectiveness of SU006668 in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of SU006668 in patients with advanced solid tumors. II. Determine the pharmacokinetics of this drug in these patients. III. Determine the objective response of patients treated with this drug. IV. Determine the toxic effects of this drug in these patients.

OUTLINE: This is a dose-escalation study. Patients receive oral SU006668 twice daily. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Cohorts of 6 to 12 patients receive escalating doses of SU006668 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 or 4 of 12 patients experience dose-limiting toxicity. Patients are followed at 30 days and then every 3 months thereafter.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of one of the following advanced malignancies: Breast Colorectal Non-small cell lung Gastric Pancreatic Renal Prostate Myeloma Failed standard therapy OR No effective standard therapy exists Measurable or evaluable disease No known CNS metastases Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Male or female Menopausal status: Not specified Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL Hepatic: Bilirubin no greater than 2.0 mg/dL AST and ALT no greater than 3 times upper limit of normal Renal: Creatinine no greater than 2 mg/dL OR Creatinine clearance at least 40 mL/min Cardiovascular: No myocardial infarction or severe/unstable angina within the past 6 months No evidence of uncompensated coronary artery disease by electrocardiogram or physical exam Other: No other malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix No insulin-dependent diabetes mellitus No non-insulin-dependent diabetes mellitus with clinical evidence of severe peripheral vascular disease or diabetic ulcers No manifestation of malabsorption due to prior surgery, GI disease, or unknown reasons No active inflammatory bowel disease No known intolerance to any excipients in the study drug formulation No other acute or chronic medical or psychiatric condition or laboratory abnormality that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior anticancer biologic or immunotherapy and recovered No prior SU006668 No other concurrent immunotherapy Chemotherapy: At least 4 weeks since prior anticancer chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered No concurrent chemotherapy Endocrine therapy: At least 4 weeks since prior hormonal therapy No concurrent hormonal therapy except for hormonal contraception or appetite stimulation Radiotherapy: Recovered from prior radiotherapy Surgery: At least 6 weeks since prior surgery At least 6 months since prior coronary/peripheral artery bypass graft surgery Prior major GI surgery allowed if no residual syptomatic manifestation of malabsorption No prior organ transplantation Other: At least 4 weeks since prior investigational agents No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Lee S. Rosen, MD, Study Chair — Jonsson Comprehensive Cancer Center